CLINICAL TRIAL: NCT06959004
Title: Substance P-Induced Migraine Attacks Without Aura: A Randomized Clinical Trial
Brief Title: Substance P-Induced Migraine Attacks Without Aura
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Haidar Al-Khazali, Sub-Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-23034165
Record Dates: First submitted 2025-05-05; First posted 2025-05-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Migraine
Keywords: Headache; Migraine; Pain; Substance P
MeSH Terms: conditions — Migraine Disorders; Headache; Pain | interventions — Substance P

STUDY DESIGN:
Intervention Model Description: This single-center trial applies a randomized, double-blind, placebo-controlled, two-way crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Substance P (Experimental): Substance P will be administered by intravenous infusion.
  Interventions: Drug: Substance P
- Placebo (Placebo Comparator): Placebo (isotonic saline) will be administered by intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Substance P — The participants will receive a continuous intravenous infusion of 20 mL of substance P (4.0 pmol/kg/min) over 20 minutes.
  Arms: Substance P
Drug: Placebo — The participants will receive a continuous intravenous infusion of 20 mL of placebo (isotonic saline) over 20 minutes.
  Arms: Placebo

SUMMARY:
Substance P is a neuropeptide implicated in the pathogenesis of headache. This study investigates whether its administration can trigger migraine attacks in individuals with migraine without aura.

DETAILED DESCRIPTION:
Substance P is a vasoactive neuropeptide of the tachykinin family, expressed in various cell types, including primary afferents of the trigeminal ganglion that innervate the meninges and associated vasculature. Its most well-established role is in nociceptive signaling, and accumulating evidence implicates substance P in the pathogenesis of headache. This study investigates whether intravenous infusion of substance P can induce migraine attacks in individuals with a history of migraine without aura. To test this, the investigators will conduct a randomized, double-blind, placebo-controlled, two-way crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age upon entry into screening
* A body weight of 50 to 100 kg
* History of migraine without aura for ≥12 months and in accordance with ICHD-3
* Between 1-5 monthly migraine days without aura on average across the 3 months prior to screening

Exclusion Criteria:

* Any history of a primary or secondary headache disorder other than migraine without aura and infrequent episodic tension-type headache
* Any history of moderate to severe traumatic brain injury
* Any history of cardiovascular disease, including cerebrovascular diseases
* Any history of pulmonary disease
* Any other clinically significant disorders, conditions, or diseases that might impact the safety of the subject or interfere with the study's evaluation, procedures, or completion, aside from those mentioned above. This includes any relevant medical history or evidence that, in the opinion of the site investigator, might pose a risk to the subject or impact the validity of the study results
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior
* Female subjects of childbearing potential with a positive pregnancy test during any study visit
* Cardiovascular disease of any kind, including cerebrovascular diseases
* Hypertension (systolic blood pressure of ≥150 mmHg and/or diastolic blood pressure of ≥100 mmHg) prior to the start of infusion on the experimental day
* Hypotension (systolic blood pressure of ≤90 mmHg and/or diastolic blood pressure of ≤50 mmHg)
* Daily use of any medication other than contraceptives
* Intake of any medication other than contraceptives within 48 hours of infusion start
* Headache of any intensity within 48 hours of infusion start
* Migraine attack within 5 days of infusion start
* Aura within 48 hours of infusion start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of migraine attacks without aura | 12 hours
  The difference in the incidence of migraine attacks without aura between substance P and placebo during the 12-hour observational period after infusion start.

SECONDARY OUTCOMES:
Headache intensity scores | 12 hours
  The secondary outcome is the difference in the area under the curve (AUC) for headache intensity scores between substance P and placebo during the 12-hour observational period after infusion start.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data not published within this article will be made available on reasonable request from any qualified investigator.